CLINICAL TRIAL: NCT07246486
Title: The Composition of the Intesinal Microbiome in Women With Complication-free Pregnancy and Women With Recurrent Spontaneous Abortions.
Brief Title: Composition of the Intestinal Microbiome in Patients With Recurrent Spontaneous Abortions.
Status: Completed | Type: Observational
Sponsor: Dr. Natascha Köstlin-Gille (Other)
Collaborators: German Center for Infection Research (Other)
Responsible Party: Sponsor-Investigator, Dr. Natascha Köstlin-Gille, PD Dr. med. Natascha Köstlin-Gille, University Hospital Tuebingen
Organization: University Hospital Tuebingen (Other)
Other Study IDs: 730/2020BO2
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2020-11

CONDITIONS: Spontaneous Abortion
Keywords: microbiome, spontaneous abortion
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples for microbiome analyses Bloodserum and urine for hormone levels for bacterial metabolic products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 2 spontaneous abortions: non-pregnant women with two spontaneous abortions in medical history
- 3 spontaneos abortions: non-pregnant women with two spontaneous abortions in medical history
- controle-group: non-pregnant women with at least one complication-free pregnancy with no premature birth or late abortion in medical history

SUMMARY:
Up to 50% of all women suffer of a spontaneous abortion. Having two/three or more spontaneous abortions is one of the main reasons of unwanted childlessness. It is well known that the intestinal microbiome has many important roles in a healthy organism. Simultaneously, a dysbiosis can lead to diseases like, for example, chronic inflammatory bowel diseases, autoimmune diseases or diabetes. Several studies showed that there is a connection between a vaginal dysbiosis and premature birth or late abortion. It is still unclear what effects the composition of the intestinal microbiome before pregnancy has on the course of pregnancy.

This study will be investigate if there is a connection between the composition of the intestinal microbiome and the occurence of recurrent spontaneous abortions.

DETAILED DESCRIPTION:
This study wants to investigate if there is a connection between the composition of the intestinal microbiome before pregnancy and the occurence of recurrent spontaneous abortions. Herefore samples of stool and blood serum will be sampled from patients with 2 or 3 consecutive spontaneous abortions and from patients with no abortions or premature birth and at least one pregnancy without complications. Microbiome analyses will be performed on the stool samples, the bloodserum will be used to analyze bacterial metabolic products.

In this study 60 non-pregnant women will be included. 20 women with at least one complication-free pregnancy and no abortions or premature birth in medical history and 40 non-pregnant women with two or three recurrent spontaneous abortions in medical history.

ELIGIBILITY:
Inclusion Criteria:

* Patient of the fertility center of the university hospital Tübingen
* 2 or 3 spontaneous abortions in medical history

Exclusion Criteria:

* Age under 18 years, age over 40 years
* Current pregnancy
* Immunosuppressive therapy
* Antibiotic therapy up to four weeks before admission
* Acute infection
* Orale intake of probiotics up to four weeks before admission

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: non-pregnant women between 18 and 40 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Intestinal microbiome | 48 month
  Microbiome Analysis from the stool samples
Hormon levels | 48 month
  Hormone levels of Estrogen, Progesterone from blood and urine samples
bacterial metabolic products | 48 month
  Metabolic products phytoestrogene enterodiol, enterolactone from blood and urine samples

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided